CLINICAL TRIAL: NCT06073782
Title: The Effect of Patient Education and Text Message Reminders on Bowel Preparation and Anxiety Level Before Colonoscopy
Brief Title: Patient Education and Text Message Reminders in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Arif Murat Alagöz, Arif Murat Alagöz, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-MA-292
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Colon Disease; Educational Problems
Keywords: colonoscopy; patient education
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education Group (Experimental): The training material will be created by researchers by reviewing national and international guidelines for colonoscopy practices. Using the "Colonoscopy Patient Preparation Guide", individuals will be given face-to-face, information and preparation training on colonoscopy preparation, its importance, the preparation medication to be used and the procedure process for an average of 15-20 minutes in a private room in the unit. After the training, individuals will be given the "Colonoscopy Patient Preparation Guide" brochure developed by the researchers.
  Interventions: Other: Education Group
- Text Message Group (Experimental): Individuals will be subjected to the routine colonoscopy preparation procedure of the hospital by the investigator. Starting three days before the colonoscopy is performed, individuals will be informed via text messages about the foods and beverages that they can consume in their diet and those that are forbidden to consume until the morning of the colonoscopy, the amount of fluids they should consume daily, the use of medication, the use of soda and enema, appointment time reminders.
  Interventions: Other: Text Message Group
- Control Group: (No Intervention): Individuals in the control group will be subjected to the standard procedure applied in the clinic. No additional education and educational brochures will be given to these patients and text message reminders will not be applied.

INTERVENTIONS:
Other: Education Group — The training material will be created by researchers by reviewing national and international guidelines for colonoscopy practices. Using the "Colonoscopy Patient Preparation Guide", individuals will be given face-to-face, information and preparation training on colonoscopy preparation, its importance, the preparation medication to be used and the procedure process for an average of 15-20 minutes in a private room in the unit.
  Arms: Education Group
Other: Text Message Group — . Starting three days before the colonoscopy is performed, individuals will be informed via text messages about the foods and beverages that they can consume in their diet and those that are forbidden to consume until the morning of the colonoscopy, the amount of fluids they should consume daily, the use of medication, the use of soda and enema, appointment time reminders.
  Arms: Text Message Group

SUMMARY:
This study will be conducted to examine the effects of detailed education and text message reminders given to patients undergoing colonoscopy on bowel cleansing, vital signs and anxiety.

DETAILED DESCRIPTION:
İntroduction: The highest level of bowel preparation before the colonoscopy procedure is necessary for the successful completion of colonoscopy. Considering that the bowel preparation procedures required for colonoscopy are performed by patients, it is very important to inform patients about the content and duration of diet and bowel preparation practices. Today, with the widespread use of technology in our lives, technological education methods such as web-based trainings, text message reminders, telemedicine methods have started to be used in patient education methods as well as classical methods.

Purpose: This study will be conducted to examine the effects of detailed education and text message reminders given to patients undergoing colonoscopy on bowel cleansing, vital signs and anxiety.

Method: This study will be a randomized controlled trial. hospital. The sample of the study will include individuals who will undergo colonoscopy procedure in the endoscopy unit of a state hospital and who meet the inclusion criteria. Data will be collected using personal information form, beck anxiety scale, boston bowel readiness scale. In this study, in addition to the standard patient education protocol, the effectiveness of colonoscopy education with more intensive content and supported by visuals and diagrams will be evaluated in the education group. Individuals in the other group will receive text message reminders, which is one of the new methods that have started to be used in patient education with the technology that has become widespread today.

Conclusion: It is thought that more intensive and materialized trainings and text message reminders to patients compared to standard colonoscopy preparations will increase the level of bowel cleansing, improve vital signs and reduce anxiety.

ELIGIBILITY:
Inclusion Criteria:

Individuals who understand Turkish

Individuals who know how to use a phone and read text messages

Individuals over 18 years of age

Patients undergoing colonoscopy for the first time

Exclusion Criteria:

Patients with cognitive dysfunction

Patients with neuro-psychiatric disorders

Individuals who do not know how to use a phone

Individuals undergoing colonoscopy in emergency situations

Individuals who did not give consent to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Scale | One day
  Beck Depression Scale (BDS) was developed by Beck. The scale was created to include clinical symptoms seen in depression. The items of the BDS are organized based on clinical observations and data. The scale consists of 21 symptom categories. Each symptom category is addressed with scored sentences ranging from 0-3. The maximum score that can be obtained from the scale is 63. A high total score on the scale indicates a high level or severity of depression
Boston Bowel Readiness Scale | One day
  The scale has a four-point (0-3) scoring system applied separately for each of the three parts of the colon.
  3- 0 (İnsuffıcıent) : Unprepared colon in which the mucosa cannot be evaluated due to uncleared solid fecal matter.
  1. (Bad) = Part of the mucosa is visible in the colon, but other parts are not visible due to contamination, residual fecal matter and/or opaque fluid.
  2. (Good) = Colon mucosa is well visualized but there is a small amount of impurities, small pieces of stool and/or opaque fluid.
  3. (Excellent) = The entire mucosa of the colon is well visible. No impurities, small pieces of pus or opaque fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Neşe Uysal, Study Chair — Amasya U
Locations (1):
- Amasya U, Amasya, Turkey (Türkiye)